CLINICAL TRIAL: NCT05694403
Title: Follow up of Stroke Patients by Neurologists and GP's: How Smooth is the Internal Communication and is There Room for Improvement?
Brief Title: Follow up of Stroke Patients by Neurologists and General Practitioners
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Vrije Universiteit Brussel (Other)
Responsible Party: Principal Investigator, Margaux Vanderstraeten, General practitioner in training, principal investigator, Vrije Universiteit Brussel
Other Study IDs: 22258PSFU
Record Dates: First submitted 2022-07-25; First posted 2023-01-23 (Actual); Last update posted 2023-08-14 (Actual); Status verified 2023-08

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Neurologists
  Interventions: Other: Survey
- General practitioners
  Interventions: Other: Survey

INTERVENTIONS:
Other: Survey — Questionnaire

SUMMARY:
From the region around Brussels there are currently few data on how the post-stroke process take place and how satisfied the care providers are with it. For this reason, this survey is set up with the aim of examining four pillars: the epidemiology of stroke, communication between neurologists and GPs and satisfaction with it, secondary prevention of cardiovascular disease and control/treatment of the most common sequelae after stroke. In the latter two, the emphasis is on detection and treatment, and explicitly on whose task this is (neurologist versus GP), with the aim of verifying the mutual consensus on treatment and the subsequent detection of treatment shortcomings. This study will mainly consist of interviewing general practitioners and neurologists in the periphery of Brussels. This will be done by means of partly structured questionnaires, that will be send out to the medical professionals by contact with the central umbrella organisations of neurology in the hospitals and contact with the various general practitioners' practices (directly or through the multidisciplinary meetings per region). The questionnaires will be made up in google forms, as this programme allows efficient data processing, is eas-ily understandable for every participant and as no individual patient data will be processed.

ELIGIBILITY:
Inclusion Criteria:

* Neurologist and/or general practitioner

Exclusion Criteria:

* Not actively treating stroke patients

Ages: 24 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Neurologists and general practitioners around Brussels
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2023-09-01 (Estimated); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
secondary prevention stroke: Antithrombotics | 1,5 - 2 years
  Given that the purpose of our study is not to determine which antithrombotics are started, this will not be determined. What will be asked, however, is which healthcare provider starts this and whose task this is considered to be. Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
secondary prevention stroke: Hypertension | 1,5 - 2 years
  This study will ask who starts antihypertensive drugs, whose task this is considered, how blood pressure is monitored and what the target values are. Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
secondary prevention stroke: Smoking | 1,5 - 2 years
  The questionnaire will ask whether healthcare providers themselves actively detect smoking behaviour and how this smoking behaviour is addressed. (ex. via medication, consultation with tabacologist etc) Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
secondary prevention stroke: Diabetes | 1,5 - 2 years
  The questionnaire will ask whether diabetes is actively detected by the healthcare provider himself, whether the treatment is subsequently started/adjusted himself and whose task this is according to them (neurologist, GP, diabetologist,...)
  At the end, it will also be asked whether healthcare providers would like to see changes in secondary prevention of stroke (open question, all answers will be checked) and whether the healthcare provider considers themselves to be capable enough to follow up secondary prevention in stroke patients (as this seems to be a good measure of the quality of currently available guidelines). Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
secondary prevention stroke: general | 1,5 - 2 years
  At the end, it will also be asked whether healthcare providers would like to see changes in secondary prevention of stroke (open question, all answers will be checked) and whether the healthcare provider considers themselves to be capable enough to follow up secondary prevention in stroke patients (as this seems to be a good measure of the quality of currently available guidelines). Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
sequelae of stroke: Fatigue | 1,5 - 2 years
  During the study, it will check whether fatigue is detected (example: if the treating physician often actively asks the patiënt for mental and/or physical fatigue) and what treatment is instituted. (example: psychologist, physiotherapy,...) Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
sequelae of stroke: Depression | 1,5 - 2 years
  The questionnaire will explore whether depression itself is detected by the healthcare provider, how this is done (screening questions, heteroanamnesis,...), whose job it is and whether a referral is made and to whom. Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)
sequelae of stroke: Sexual dyfunction | 1,5 - 2 years
  This study will evaluate whether sexual dysfunction is being asked, whether and what treatment is initiated. (example: medication, couples therapy etc.) Values will be reflected in ratios and percentages (%) of healthcare providers (both differences interdisciplinary and intradisciplinary)